CLINICAL TRIAL: NCT06291493
Title: Clinical Evaluation of Precision for the Potassium (K) Test in Capillary Specimens Using the i-STAT CG8+ Cartridge With the i-STAT 1 Analyzer
Brief Title: Precision Study Measuring Potassium (K) in Capillary Specimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Point of Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CS-2024-0002
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Precision of Potassium (K) Test in Capillary Whole Blood
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Capillary precision analysis will be performed for Potassium K.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Precision assessment of Potassium (K) test in capillary blood sample (Other): Prospectively collected capillary specimens from two separate fingerstick blood draws.
  Interventions: Diagnostic Test: Fingerstick blood draw

INTERVENTIONS:
Diagnostic Test: Fingerstick blood draw — Capillary blood specimen collected from two separate fingerstick blood draws.
  Other Names: Blood draw

SUMMARY:
Assessing precision of i-STAT K test using the IUO i-STAT CG8+ cartridge on the i-STAT 1 Analyzer.

DETAILED DESCRIPTION:
The objective of this study is to assess the precision of the i-STAT K test using the IUO i-STAT CG8+ cartridge on the i-STAT 1 Analyzer with investigational software using results from two (2) different fingerstick specimens from the same subject across the K measurement range.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated consent form (if required by the IRB)
* ≥ 18 years of age

Exclusion Criteria:

• Prior enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Precision for Potassium (K) Test | Up to 5 minutes
  Clinical Evaluation of Precision for the Potassium (K) Test in Capillary Specimens using the i-STAT CG8+ Cartridge with the i-STAT 1 Analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Manish Gupta, BS, MBA, Study Director — Abbott Point of Care
Locations (4):
- United States (3):
  - University of Maryland, Baltimore (UMD), Baltimore, Maryland
  - Penn State Health Milton S. Hershey Medical Center (Hershey), Hershey, Pennsylvania
  - Eastside Research Associates (ERA), Redmond, Washington
- Abbott Point of Care (APOC), Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No